CLINICAL TRIAL: NCT07147881
Title: Prospective Real-World Evidence Study of the IpsiHand® System in Adult Stroke Survivors
Status: Not yet recruiting | Type: Observational
Sponsor: Neurolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RWE_002
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Stroke; Hemiparesis After Stroke; Brain Computer Interface
Keywords: Neurolutions; IpsiHand; Stroke; Hemiparesis after stroke; BCI
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Adult stroke patients with upper extremity hemiparesis.: Chronic Stroke Patients (≥ 6 months post-stroke) age 18 or older undergoing stroke rehabilitation with use of the IpsiHand® System.
  Interventions: Device: IpsiHand

INTERVENTIONS:
Device: IpsiHand — IpsiHand is a therapeutic device that uses a brain-computer interface system which detects neural signals associated with motor intent and translates them into assisted hand movements in individuals with upper extremity impairment following a stroke.
  Other Names: IpsiHand Therapy; BCI Therapy

SUMMARY:
This study focuses on monitoring real-world customers who have been prescribed the IpsiHand® as part of their rehabilitation post-stroke. This study aims to evaluate their progress over time, assessing motor recovery, functional independence in activities of daily living (ADLs), caregiver burden, and health economic outcomes.

DETAILED DESCRIPTION:
IpsiHand® is an FDA-authorized, non-invasive, BCI-based device that is indicated for use in chronic stroke patients (≥ 6 months post stroke) age 18 or older undergoing stroke rehabilitation, to facilitate muscle re-education and for maintaining or increasing range of motion in the upper extremity. Through utilization of EEG signals from the unaffected side of the brain, the device enables stroke survivors to control a robotic hand orthosis, facilitating functional reorganization of the brain and improved motor recovery.

ELIGIBILITY:
Inclusion Criteria:

1. Adult age 18-85 years.
2. Diagnosis of stroke six or more months prior with upper extremity weakness.
3. Has received an IpsiHand® system as a commercial customer for stroke rehabilitation.

Exclusion Criteria:

1. Severe cognitive impairment that would impede utilization of IpsiHand®
2. Any contraindications to IpsiHand® device use
3. Inability to comprehend English

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Chronic stroke patients (≥ 6 months post-stroke) age 18 or older undergoing rehabilitation using the IpsiHand® System.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer - Upper Extremity (FM-UE) , Manual Long Form | Baseline visit and at 4-week, 8-week, 12-week, 16-week, 20-week, 24-week, 28-week, 32-week, 36-week, 12-months, and 24 months of IpsiHand® device use, or until completion of IpsiHand® device use if occurring prior to 24 months.
  Valid assessment tool of upper extremity motor function in persons chronic stroke with moderate to severe deficits. Lowest score 0, highest score 66.

SECONDARY OUTCOMES:
The Barthel Index | Baseline visit and at 4-week, 8-week, 12-week, 16-week, 20-week, 24-week, 28-week, 32-week, 36-week, 12-months, and 24 months of IpsiHand® device use, or until completion of IpsiHand® device use if occurring prior to 24 months.
  Assessment tool that measures a person's functional independence in activities of daily living and self-care.
Zarit Caregiver Burden Scale (ZBI) | Baseline Visit, 12-Week, 24-Week, 36 Week, 12-Months, and 24-Months post-use of IpsiHand Device or at time of completion of IpsiHand device use if occurring prior to 24-Months.
  Widely used questionnaire designed to assess the level of burden experienced by caregivers.
Patient Specific Functional Scale (PSFS) | Baseline visit and at 4-week, 8-week, 12-week, 16-week, 20-week, 24-week, 28-week, 32-week, 36-week, 12-months, and 24 months of IpsiHand® device use, or until completion of IpsiHand® device use if occurring prior to 24 months.
  patient-reported outcome measure used to assess an individual's ability to perform specific functional activities that are important to them. It is commonly used in rehabilitation and clinical settings to track progress over time in response to treatment.
Euro-QOL5D5L | Baseline Visit, 12-Week, 24-Week, 36 Week, 12-Months, and 24-Months post-use of IpsiHand Device or at time of completion of IpsiHand device use if occurring prior to 24-Months.
  Patient-reported outcome measure used to assess health-related quality of life (HRQoL) across different diseases and treatments. It is widely used in clinical research, health economics, and healthcare decision-making to quantify the impact of health conditions and interventions on daily living

CONTACTS AND LOCATIONS:
Overall Officials: Seth Wilk, PhD, Principal Investigator — Neurolutions, Inc.; Lee Fleisher, MD, Principal Investigator

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared because the dataset contains protected health information from routine clinical care. Even with de-identification, there remains a risk of re-identification, and confidentiality obligations under HIPAA and applicable privacy laws prevent sharing.

REFERENCES:
- [Background] Rustamov N, Humphries J, Carter A, Leuthardt EC. Theta-gamma coupling as a cortical biomarker of brain-computer interface-mediated motor recovery in chronic stroke. Brain Commun. 2022 May 25;4(3):fcac136. doi: 10.1093/braincomms/fcac136. eCollection 2022. PMID 35702730
- [Background] Rustamov N, Souders L, Sheehan L, Carter A, Leuthardt EC. IpsiHand Brain-Computer Interface Therapy Induces Broad Upper Extremity Motor Recovery in Chronic Stroke. medRxiv [Preprint]. 2023 Aug 28:2023.08.26.23294320. doi: 10.1101/2023.08.26.23294320. PMID 37693482
- [Background] Bundy DT, Souders L, Baranyai K, Leonard L, Schalk G, Coker R, Moran DW, Huskey T, Leuthardt EC. Contralesional Brain-Computer Interface Control of a Powered Exoskeleton for Motor Recovery in Chronic Stroke Survivors. Stroke. 2017 Jul;48(7):1908-1915. doi: 10.1161/STROKEAHA.116.016304. Epub 2017 May 26. PMID 28550098
- See also: FDA De Novo Authorization — https://www.accessdata.fda.gov/cdrh_docs/reviews/DEN200046.pdf